CLINICAL TRIAL: NCT02584569
Title: A Phase 1, Open-Label, Positron Emission Tomography Study With [18F]MNI-794 to Determine Phosphodiesterase 2A Brain Enzyme Occupancy of TAK-915 After Single-Dose Oral Administration in Healthy Subjects
Brief Title: Phase 1 TAK-915 Single-Dose Positron Emission Tomography (PET) Occupancy Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-915-1002; U1111-1168-0766 (Registry Identifier: WHO)
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Healthy Volunteers
Keywords: Drug therapy
MeSH Terms: interventions — TAK-915

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-915 (Experimental): TAK-915 100 mg suspension, orally, once on Day 1. Additional TAK-915 dose levels may be incorporated based on dose level review meetings (DLRMs) following approximately every 2 participants and based on prior occupancy, duration of occupancy, safety, tolerability, and available pharmacokinetic (PK) data.
  Interventions: Drug: TAK-915

INTERVENTIONS:
Drug: TAK-915 — TAK-915 oral suspension

SUMMARY:
This phase 1 study will be conducted to examine the degree and duration of brain PDE2A enzyme occupancy /target engagement as a function of TAK-915 plasma concentration in order to guide dosing and schedule for future clinical studies in schizophrenia with TAK-915.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-915. TAK-915 is being tested to examine the degree and duration of brain phosphodiesterase 2A (PDE2A) enzyme occupancy/target engagement as a function of TAK-915 plasma concentration in order to guide dosing and schedule for future clinical studies in schizophrenia. This study will look at PDE2A brain enzyme occupancy in the putamen as a function of TAK-915 plasma concentration, as assessed using the positron emission tomography (PET) ligand [18F]MNI-794 after single dosing of TAK-915.

The study will enroll approximately 16 patients in total and within that total, allow up to 5 dose levels and up to 6 subjects per dose level. All participants will receive a single dose of TAK-915 on Day 1. The initial TAK-915 dose level to be studied is 100 mg. Subsequent dose levels may be lower or higher and will be determined through dose level review meetings (DLRMs) following approximately every 2 participants and based on prior occupancy, duration of occupancy, safety, tolerability, and available pharmacokinetic (PK) data.

This single center trial will be conducted in the United States. The overall time to participate in this study is up to 55 days. Participants will make multiple visits to the clinic, and will be contacted by telephone 22 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Is a healthy male, or female of non-childbearing potential, aged between 18 and 55 years, inclusive.
2. Weighs at least 45 kg and has a body mass index (BMI) between 18.0 and 30.0 kg/m^2.

Exclusion Criteria:

1. Has a known history or evidence of a clinically significant disorder (including neurologic and psychiatric) or disease that in the opinion of the study investigator would pose a risk to the participant's safety or interfere with the study evaluation, procedures, or completion.
2. Contraindication to magnetic resonance imaging (MRI) based on the standard MRI screening questionnaire.
3. Have had exposure to any radiation >15 millisievert (mSv)/year (eg, occupational or radiation therapy) within the previous year prior to Baseline imaging.
4. Has a known hypersensitivity to any component of the formulation of TAK-915 or related compounds, or to [18F]MNI-794 or to any of its components.
5. Clinically significant abnormal findings on brain MRI scan or findings on brain MRI that may interfere with the interpretation of the positron emission tomography (PET) imaging.
6. Use of any herbal or prescription medications within 30 days prior to Baseline Imaging Check-in; use of any over-the-counter medications or vitamin supplements within 7 days prior to Baseline Imaging Check-in.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Phosphodiesterase 2A (PDE2A) Brain Enzyme Occupancy in the Putamen as a Function of TAK-915 Plasma Concentration for each subject | 2 PET scans occurring on Day 1 or 1 PET scan on Day 1 and 1 on Day 2.
  Assessed for each subject using the PET ligand [18F]MNI-794 after single dosing of TAK-915, obtained from non-displaceable binding potential (BPnd).

SECONDARY OUTCOMES:
Plasma PK concentrations for each subject post tracer injection for each PET scan period following TAK-915 dosing | t=0, t=45 min and t=90 min (after tracer injection) during each PET scan period.
Dose and exposure of TAK-915 that correspond to PDE2A occupancy in the putamen of at least 45%. | At multiple time points (up to 90 minutes after tracer injection) during each PET scan period.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (1):
- New Haven, Connecticut, United States